CLINICAL TRIAL: NCT01618981
Title: LEft Atrial Pacing in Diastolic Heart Failure
Acronym: LEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LAURENT PHRC N 2011
Record Dates: First submitted 2012-06-07; First posted 2012-06-14 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Atrial Dyssynchrony Syndrome; Left Atrio-ventricular Asynchrony
Keywords: Heart failure with preserved ejection fraction; atrial dyssynchrony syndrome; left atrio-ventricular asynchrony; pacemaker; left atrial pacing therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- first active (Experimental)
  Interventions: Procedure: pace make active/inactive cross over
- first inactive (Experimental)
  Interventions: Procedure: pace make active/inactive cross over

INTERVENTIONS:
Procedure: pace make active/inactive cross over

SUMMARY:
The purpose of this study is to assess left atrial pacing therapy in patients with atrial dyssynchrony syndrome and heart failure with preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Sinus rhythm, PR < 220ms, QRS < 110ms
* Heart failure (NYHA class III-IV or II with hospitalization for heart failure)
* Ejection Fraction > 50%, restrictive mitral inflow, Lateral E/e' > 12 or septal E/e' > 15, Left atrial index volume > 34 ml/m²
* Atrial dyssynchrony syndrome: (TTE) inter-atrial time delay ≥ 70ms (difference between tricuspid and mitral P-A intervals or between mitral and tricupsid P-A' intervals with DTI)
* Left atrio-ventricular asynchrony: Time Difference between tricupsid and mitral A wave duration ≥ 35ms.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2012-11 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France